CLINICAL TRIAL: NCT06216834
Title: Quality of Life and Psychosocial Status of Young-onset Patients With Rectal Cancer After Surgery: a Cross-sectional Muti-questionnaire Survey
Brief Title: Quality of Life and Psychosocial Status of Young-onset Patients With Rectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Teng Qiong, Resident physician, Shandong Provincial Hospital
Other Study IDs: SWYX:NO.2023-546
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Rectal Cancer
Keywords: Young-onset rectal cancer; Quality of life; Psychosocial status; Muti-questionnaire
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Colorectal cancer is one of the leading cancers worldwide. Although the majority of CRC cases are typically diagnosed in individuals older than 50 years of age, recent international studies have highlighted the importance of younger adults (< 50) are gradually increasing. Young cancer survivors often have poorer quality of life, disrupted social and sexual health, and increased mental health-related risks such as depression and anxiety. Especially for patients with rectal cancer, patients may suffer from sexual dysfunction, urinary system problems and loss of normal bowel function after radical resection of rectal tumors, and some patients may also need to undergo ostomy, which may have adverse effects on the quality of life and mental health of patients after surgery. Given that the incidence of colorectal cancer in young adults continues to rise worldwide, there is a need to better understand the impact of this particular disease on postoperative quality of life in young adults. This study intends to retrospectively analyze the clinical characteristics of the patients, and further summarize the impact of rectal cancer surgery on the quality of life of patients through follow-up.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common malignancy worldwide and the second leading cause of cancer death. The incidence of CRC has remained stable or declined in high-income countries over the past decade, possibly due to a series of screening and prevention measures aimed at people aged 50-70 years. However, there is an increased incidence of rectal cancer in people younger than 50 years of age, which is known as young-onset RC (YO-RC). By 2030, YO-RC is expected to account for 23% of rectal cancers. In America, the proportion of people under 55 years of age newly diagnosed has increased from 11% in 1995 to 20% in 2019, and the incidence of RC in people under 50 years of age has increased by about 2% per year. Due to the early detection of routine physical examination, advances in imaging, improved surgical techniques, and advances in chemoradiotherapy, colorectal cancer mortality is on a downward trend, with overall mortality declining by 57% from 1970 to 2020. Therefore, those who are diagnosed with RC under the age of 50 are also called young-onset rectal cancer (YO-RC). Prognostic analyses of YO-RC have been mixed, with some studies suggesting worse survival outcomes in younger patients, while others have shown no difference between younger and older patients. In view of the difficulty of curing cancer and its complexity, traditional evaluation indicators such as survival time, remission period, treatment-related toxicity and tumor remission rate cannot comprehensively and accurately evaluate the medical outcome of cancer patients. More and more people pay attention to the QOL of patients after treatment, which can comprehensively, objectively and truly evaluate the medical outcome from the perspective of patients. Surgery is the basis of curative treatment for RC. Problems that arise after RC surgery can impair quality of life (QOL), such as fatigue, abdominal pain, changes in bowel function, and decreased sexual function. In addition, postoperative radiotherapy and chemotherapy can also reduce patients' QOL. It is important to note that YO-RC patients may experience very different psychosocial status (PS) than older patients, with mental health issues such as anxiety and depression being more prominent. At the same time, because YO-RC patients have higher requirements for postoperative QOL, it is necessary to adopt standardized quantitative scales to measure the postoperative situation of this group of people, so that clinicians can provide more effective interventions. Here, we used the questionnaires, developed by the European Organization for Research and Treatment of Cancer (EORTC), to assess the QOL of patients with CRC. Several standardized psychological and functional scales (previously applied to studies of other post-surgical tumors) were used to assess mental stress, body image anxiety, and work ability in patients after RC surgery. This study is the first to evaluate the five-year QOL and PS in YO-RC patients after surgery using multiple questionnaires. Based on our research results, the QOL and PS of patients can be better predicted, and then timely measures can be taken to help patients improve the QOL and relieve psychological pressure.

ELIGIBILITY:
Inclusion Criteria:

* 1. Preoperative colonoscopy and pathological examination were performed to confirm the pathological diagnosis of rectal cancer; 2. Abdominal and pelvic CT examination and MRI examination were performed before operation to carefully evaluate the extent of tumor invasion and whether there was distant metastasis. 3. The patient's clinical data (contact information, age, gender, hospitalization record, colonoscopy report, postoperative pathological report, operation record, informed consent) were recorded comprehensively; 4. Patients with R0 resection; 5. The patients are more than 18 years old and less than 50 years old.

Exclusion Criteria:

* 1. Patients with other malignant tumors; 2. Previous history of other malignant tumors; 3. Patients with inflammatory gastrointestinal disease; 4. Emergency surgery; 4. Patients with preoperative mental illness or cognitive impairment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young patients undergoing radical resection for rectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Quality-of-life scores | From September 2023 to September 2024
  patients' quality of life after surgery
psychosocial status | From September 2023 to September 2024
  patients' psychosocial status after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China